CLINICAL TRIAL: NCT06831409
Title: Using CTA Measures to Define Cardiac Risk In NFL Alumni
Acronym: GAMEFILM
Status: Recruiting | Type: Observational
Sponsor: HeartFlow, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 11072024
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease (CAD); Heart Disease; Coronary Atherosclerosis
Keywords: NFL; Heart Disease
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- NFL Alumni: A retired NFL player is defined as any former player who made either a practice squad or an active NFL roster.
  Interventions: Diagnostic Test: Coronary computed tomography angiography

INTERVENTIONS:
Diagnostic Test: Coronary computed tomography angiography — Coronary Computed Tomography Angiography (CCTA) is a non-invasive medical imaging test that uses X-rays to create detailed 3D images of the heart and its blood vessels, specifically the coronary arteries.

SUMMARY:
The GAMEFILM Registry is a post-market, multi-center, data collection study assessing the presence of CAD in NFL alumni.

DETAILED DESCRIPTION:
The GAMEFILM Registry is a post-market, multi-center, data collection study assessing the prevalence and severity of CAD in NFL alumni. A retired NFL player is defined as any former player who made either a practice squad or an active NFL roster. Approximately 300 participants will be included from approximately 20 sites in the US.

ELIGIBILITY:
Inclusion Criteria:

* Retired NFL player

Exclusion Criteria:

* CCTA not successfully processed for FFRct and AI-Plaque

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population is retired NFL alumni. A retired NFL player is defined as any former player who made either a practice squad or an active NFL roster.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Participants with CAD | 24 hours from the time CCTA was taken
  The proportion of participants with coronary artery disease demonstrated on coronary computed tomography angiography (CCTA).

SECONDARY OUTCOMES:
Participants with physiologically significant CAD | 24 hours from the time CCTA was taken
  1. The proportion of participants with physiologically significant CAD (FFRct ≤ 0.80)
Participants with high coronary plaque burden | 24 hours from the time CCTA was taken
  2. The proportion of participants with high coronary plaque burden (>75th percentile for age- and sex-matched peers)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Boone, Principal Investigator — Boone Heart Institute
Locations (1):
- Boone Heart Institute, Greenwood Village, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided